CLINICAL TRIAL: NCT06250959
Title: Comparing the Efficacy and Safety of Reduced-dose Chemotherapy Followed by Blinatumomab Versus hyperCVAD as Induction Therapy for Newly Diagnosed Ph-negative B-ALL: a Multicenter, Radomized, Phase 2 Study
Brief Title: RDC-Blinatumomab Versus hyperCVAD for Ph-negative B-ALL.
Acronym: BEAT-ALL-2024
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Chen Suning (Other)
Responsible Party: Sponsor-Investigator, Chen Suning, Physician, The First Affiliated Hospital of Soochow University
Organization: The First Affiliated Hospital of Soochow University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BEAT-ALL-2024
Record Dates: First submitted 2024-02-01; First posted 2024-02-09 (Actual); Last update posted 2024-04-04 (Actual); Status verified 2024-04

CONDITIONS: ALL, Adult; Philadelphia-Negative ALL
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — blinatumomab; Doxorubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Reduced-dose Chemotherapy Followed by Blinatumomab (Experimental): Reduced-dose Chemotherapy(including 1 dose of Idarubicin 8 mg/m2, 1 dose of Vincristine 1.4 mg/m2[max 2mg], and 7 days of Dexamethasone 9 mg/m2/d) followed by 2 weeks of Blinatumomab (9 ug/d d8-14, 28 ug/d d15-21) immediately. If not achieved CR/CRi, Blinatumomab 28 ug for another 14 days should be continued.
  Interventions: Drug: Blinatumomab Injection [Blincyto]
- hyperCVAD (Active Comparator): CTX 300mg/m2 q12h D1-3 VCR 1.4mg/m2 (max 2mg) D4,D11 DNR 50mg/m2, D4 DEX 40mg/d D1-4, D11-14
  Interventions: Drug: Doxorubicin

INTERVENTIONS:
Drug: Blinatumomab Injection [Blincyto] — Reduced-intensity chemotherapy followed by Blinatumomab
  Arms: Reduced-dose Chemotherapy Followed by Blinatumomab
Drug: Doxorubicin — HyperCVAD regimen
  Arms: hyperCVAD

SUMMARY:
In this study, newly diagnosed non-elderly patients with Philadelphia chromosomal negative (PH-) B-ALL were enrolled and 1:1 randomised into Reduced-intensity chemotherapy followed by Blinatumomab cohort or hyperCVAD cohort as induction therapy. The clinical remission rate, MRD negative rate and treaty-related adverse reactions were evaluated.

DETAILED DESCRIPTION:
Blinatumomab, a CD3/CD19 bisespecific T-cell conjugative antibody, has shown high efficacy in phase I/II studies of relapsed/refractory B-lymphoblastic leukemia (B-ALL), particularly in the context of low tumor burden.Meanwhile, Blinatumomab also plays an important role in rapid and efficient clearance of MRD in patients. Therefore, its use in combination with less intensive chemotherapy for initial induction therapy in newly diagnosed patients may result in favorable response rates, greater depth of remission, and lower treatment-related toxic effects.

In this study, newly diagnosed non-elderly patients with Philadelphia chromosomal negative (PH-) B-ALL were enrolled and 1:1 randomised into Reduced-intensity chemotherapy followed by Blinatumomab cohort or hyperCVAD cohort as induction therapy. The clinical remission rate, MRD negative rate and treaty-related adverse reactions were evaluated.

The regimen of consolidation therapy is recommended as multidrug combination chemotherapy (including high-dose Methotrexate or Cytarabine combined with Asparaginase) or alternating with Blinatumomab (28 ug/d×28d). If Allogeneic Hematopoietic Stem Cell Transplantation (Allo-HSCT) is not performed, consolidation therapy needs at least 4 courses before 2 years maintenance therapy.

ELIGIBILITY:
Inclusion Criteria:

* Age 15-65
* Ph-(BCR-ABL1 negative)B-ALL was diagnosed according to WHO diagnostic criteria
* Newly diagnosed patients without prior induction therapy (except hydroxyurea and glucocorticoids ≦5 days
* ECOG score 0-3
* Liver function: total bilirubin ≦ 3 times the upper limit of normal; Alanine ·aminotransferase ≦ 3 times upper limit of normal motion; Aspartate aminotransferase ≦ 3 times upper limit of normal motion; (except considering leukemia infiltration)
* Renal function: endogenous creatinine clearance ≧30ml/min
* Patients must be able to understand and willing to participate in the study and must sign the informed consent form.

Exclusion Criteria:

* Ph+ (BCR-ABL1 positive) ALL
* T cells ALL
* Mature B-cell leukemia/lymphoma, B-cell lymphoma, with extramedullary disease
* Acute mixed-cell leukemia
* Central nervous system leukemia
* HIV infection
* HBV-DNA or HCV-RNA positive
* Patients with grade 2 or higher heart failure and other patients deemed inappropriate for inclusion by the investigator
* Pregnant or breastfeeding patients
* The study patient was refused enrollment

Ages: 15 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 124 (Estimated)
Dates: Start 2024-02-05 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Composite complete remission rate | Induction therapy phase: The time of bone marrow evaluation is day 28±7.
  CR/CRi

SECONDARY OUTCOMES:
The negative rate of minimal residual lesion (MRD) | Induction therapy phase: The time of bone marrow evaluation is day 28 ±7.
  The negative rate of minimal residual lesion (MRD) during induction therapy (The threshold is 1×10^-4)
Treatment-related AE | Induction therapy phase
  Incidence of treatment-related adverse events, including severe bleeding, infection, drug-related adverse events, and organ dysfunction.
Quality of survival of patients in the induction therapy phase | Induction therapy phase
  QLQ-C30 Survival Quality Scale
Progression-free survival（PFS） | 1 year after study completion
  The time from random assignment in a clinical trial to disease progression or death from any cause.
Overall survival (OS) | 1 year after study completion
  From the time of enrollment in the study to the time of death from any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Jing Lu, MD, Principal Investigator — Soochow U
Locations (1):
- The First Affiliated Hospital of Soochow University, Suzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Yes
Study Protocol, Basic Statistical Analysis
Supporting Information: Study Protocol
Time Frame: 1 year after the publication of the summary paper